CLINICAL TRIAL: NCT05769478
Title: A Proof of Concept Study of the Effect of Amifampridine (Firdapse®) on Neuromuscular Transmission in Patients Treated With OnabotulinumtoxinA (Botox®, BTX-A)
Brief Title: Effect of Amifampridine on Neuromuscular Transmission in Patients Treated With OnabotulinumtoxinA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00091315
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-03

CONDITIONS: Botulism; Iatrogenic Botulism
Keywords: botulinum toxin injections; Systemic botulism; neuromuscular transmission; single fiber electromyography; amifampridine
MeSH Terms: conditions — Botulism | interventions — Amifampridine

STUDY DESIGN:
Intervention Model Description: before-after study that will measure neuromuscular jitter before and after administration of amifampridine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amifampridine will be orally administered to study participants (Experimental): Amifampridine will be orally administered to study participants following completion of the baseline SFEMG. Post-dose SFEMG will commence at 30 minutes following dosing and will be completed within 30 minutes. The participant will remain under observation in the Diagnostic Neurology suite for 2 hours after dosing so it is estimated that the entire protocol including monitoring will be completed within 2-3 hours.
  Interventions: Drug: Amifampridine

INTERVENTIONS:
Drug: Amifampridine — a single dose of amifampridine (20mg) will be orally administered
  Other Names: Firdapse

SUMMARY:
if amifampridine can improve neuromuscular transmission in muscles previously injected with OnabotulinumtoxinA (BTX-A)

DETAILED DESCRIPTION:
Amifampridine may also be effective in treating the sequelae of botulinum toxin injections and this study will determine if neuromuscular transmission as measured by single fiber electromyography is improved in patients treated with BTX-A following administration of amifampridine

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years of either gender and of any racial background
* Underwent BTX-A injection of facial muscles including frontalis with a total dose between 100-200 units between 80 and 150 days prior to study
* Have decision-making capacity to provide informed consent to study drug dosing and Single Fiber Electromyography (SFEMG)

Exclusion Criteria:

* History of cardiac arrhythmia
* History of seizures or uncontrolled asthma
* History of renal or hepatic disease
* History of any generalized neuromuscular disease
* History of Bell's Palsy or facial nerve trauma
* History of treatment with or sensitivity to amifampridine, 3,4 diaminopyridine (DAP) or 4-aminopyridine (Ampyra®)
* Currently experiencing sequelae of previous BTX-A treatment
* Current use of pyridostigmine (known to alter neuromuscular transmission)
* Use of any investigational drug or device within 30 days of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Percentage of abnormal pairs | Hour 3
  Wilcoxon's test for paired data will be used to analyze baseline and post-treatment percent abnormal pairs
Percentage of Jitter | Hour 3
  Wilcoxon's test for paired data will be used to analyze baseline and post-treatment mean jitter
Percentage of pairs that show blocking | Hour 3
  Wilcoxon's test for paired data will be used to analyze baseline and post-treatment percent blocking

CONTACTS AND LOCATIONS:
Overall Officials: James B Caress, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT05769478/ICF_000.pdf